CLINICAL TRIAL: NCT04766138
Title: Neurophysiological Mechanism in Sacral Neuromodulation in Patients Suffering From Fecal Incontinence
Brief Title: Trial to Evaluate Fecobionics in Healthy Subjects and Patients
Acronym: NORMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The California Medical Innovations Institute, Inc. (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Hans Gregersen, PhD, Research Professor, The California Medical Innovations Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CALMI-CLIN-2019-01
Record Dates: First submitted 2020-08-02; First posted 2021-02-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Normal Subjects; Fecal Incontinence
Keywords: anorectal; Fecobionics; defecation; bionics
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecobionics studies (Experimental): Single-arm study
  Interventions: Device: Fecobionics
- Feco BFT (Active Comparator): In this ARM Fecobionics will be used as a BFT tool
  Interventions: Device: Fecobionics

INTERVENTIONS:
Device: Fecobionics — Fecobionics is a new device to be inserted through the anal canal into rectum for studying defecation

SUMMARY:
Fecobionics combines several existing tests to provide novel insight into anorectal function. The purpose for the development was to overcome the technological controversies and disagreement between various tests and unphysiological test conditions. The aim was to imitate defecation as much as possible to the natural process. Fecobionics was developed to simulate stool and to provide the driving pressure and resulting deformations of stool along with a measure of an objective anorectal angle during defecation in a single examination. Fecobionics makes it possible to describe objectively, without disturbing the defecation process, the opening characteristics and pressure signatures during initial entry into the relaxing anal canal.

The overall goal is to provide mechanistic understanding of defecation in health and defecatory disorders. It exceeds previous attempts to make artificial stool for evaluation of defecation and integrates other technologies as well. It was designed to have a consistency and deformability of Type 4 (range type 3-5) on the Bristol stool form scale. The range from types 3-5 is found in 70% of healthy subjects. A major novelty is that Fecobionics measures pressures in axial direction; i.e., in the flow direction. It is anticipated that Fecobionics will shed light on the neurophysiology of defecation in health and disease, including understanding the effect of biofeedback and neuromodulatory effect of SNS. It will be of great value to provide endpoints in normal subjects that in future studies can be objective measures for monitoring treatment efficacy. The present protocol is on normal subjects only.

DETAILED DESCRIPTION:
Fecal continence is maintained by several mechanisms including anatomical factors, anorectal sensation, rectal compliance, stool consistency, anal muscle strength, mobility, and psychological factors. The homeostatic balance is easily disturbed by functional or structural anorectal disturbances that may coexist. Common anorectal disorders are fecal incontinence, functional anorectal pain, and functional defecation disorders. These conditions greatly affect life quality for the patients. Current technologies for anorectal functional assessment studies have limitations and often overlap is found between patient groups with lack of correlation between measurements and symptoms. Defecation physiology has been studied for many years but the mechanics and mechanosensation of defecation are still not well understood.

Fecobionics combines several existing tests to provide novel insight into anorectal function. The purpose for the development of Fecobionics was to overcome the technological controversies and disagreement between various tests and unphysiological test conditions. The aim was to imitate defecation as close as possible to the natural process. Fecobionics was developed to simulate stool and to provide the driving pressure and resulting deformations of stool along with a measure of an objective anorectal angle during defecation in a single examination. Fecobionics makes it possible to describe objectively, without disturbing the defecation process, the opening characteristics and pressure signatures during initial entry into the relaxing anal canal as well as other parameters

The overall goal is to provide mechanistic understanding of defecation in health and defecatory disorders. Fecobionics exceeds previous attempts to make artificial stool for evaluation of defecation and integrates other technologies as well. It was designed to have a consistency and deformability of Type 4 (range type 3-5) on the Bristol stool form scale. The range from types 3-5 is found in 70% of healthy subjects. A major novelty is that Fecobionics measures pressures in axial direction; i.e., in the flow direction. It is anticipated that Fecobionics will shed light on the neurophysiology of defecation in health and disease, including understanding the effect of biofeedback and neuromodulatory effect of SNS. It will be of great value to provide endpoints in normal subjects that in future studies can be objective measures for monitoring treatment efficacy. The present protocol is on normal subjects only, i.e. studying mechanisms of defecation.

ELIGIBILITY:
For Normal Subjects (in California Medical Innovations Institute):

Inclusion Criteria:

1. Subject must provide written informed consent;
2. Age 18 years and of age of legal consent;
3. Normal defecation pattern;
4. Within normal range for fecal incontinence severity index (FISI) and Wexner Constipation Scoring System (CSS) scores.

Exclusion Criteria:

1. Female, who is pregnant or lactating;
2. Prior abdominal surgery;
3. Diagnosis of fecal incontinence, constipation or anorectal pain.

For Patients with Fecal Incontinence (in University of California, San Diego):

Inclusion Criteria:

1. Subject must provide written informed consent;
2. Age 18 years and of age of legal consent;
3. Diagnosed Fecal Incontinence and scheduled for sacral neuromodulation treatment

Exclusion Criteria:

1. Female, who is pregnant or lactating;
2. Prior abdominal surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Duration-based device expulsion parameters | 1 year
  Expulsion Duration - The time it takes to defecate Fecobionics
Pressure-based device expulsion parameters | 1 year
  Pressure difference between front and rear of Fecobionics device - A measure of anal sphincter relaxation and key to the determination of defecation phases. Pressure profiles

SECONDARY OUTCOMES:
Mechanical-based expulsion parameters Endpoints | 1 year
  Mechanical Tension of Fecobionics Device (Pressure multiplied with radius).
Device orientation and bending-based expulsion parameters | 1 year
  orientation of the device (degrees) and bending angle (degrees, a proxy of the anorectal angle during defecation)
Shape-based expulsion parameters | 1 year
  bag shape during defecation. Topographic characteristics of Fecobionics.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gregersen, PhD, Principal Investigator — California Medical Innovations Institute
Locations (1):
- California Medical Innovations Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No